CLINICAL TRIAL: NCT02504294
Title: The Pieda Study: A Phase 3b Investigation Of Erythropoietin Drugs Using A Specified Dosing Algorithm: A Randomized Open Label Dosing Study In Adult Chronic Kidney Disease Subjects On Hemodialysis
Brief Title: A Phase 3b Study of Erythropoietin Drugs Using a Specified Dosing Algorithm in Patients With Chronic Kidney Disease on Hemodialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ZIN-EPO-1503; C3461008 (Other: Alias Study Number)
Record Dates: First submitted 2015-07-20; First posted 2015-07-21 (Estimated); Results first posted 2018-06-13 (Actual); Last update posted 2018-06-13 (Actual); Status verified 2018-05

CONDITIONS: Chronic Kidney Disease (CKD)
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — ferryl iron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Epoetin Hospira (Other): Epoetin Hospira Arm
  Interventions: Biological: Epoetin Hospira Arm; Drug: IV Iron
- Standard of Care (Other): Standard of care arm
  Interventions: Other: Standard of Care Arm; Drug: IV Iron

INTERVENTIONS:
Biological: Epoetin Hospira Arm — Epoetin Hospira Arm: Epoetin Hospira will be administered intravenously (IV) per the analogous version of the Fresenius Medical Care North America (FMCNA) cMAB 1 (inclusive of version 1.0, 1.1,...)erythropoietin stimulating agents (ESA) dosing algorithm for Epoetin Hospira for 24 weeks. Subjects will have Epoetin Hospira initiated using the same ESA dose level and frequency of administration for Epogen prior to randomization into the trial. Subjects will also receive IV iron per the FMCNA protocol that is standard of care at FMCNA clinics.
  Arms: Epoetin Hospira
Other: Standard of Care Arm — Standard of care arm: No interventions will be performed in this arm for the clinical study; and subjects will receive ongoing standard of care, which includes Epogen administered IV per the FMCNA cMAB 5 (inclusive of versions 5.0, 5.1,....) ESA dosing algorithm and IV iron per the FMCNA protocol that is standard of care, at FMCNA clinics during the contemporaneous 24 week period.
  Arms: Standard of Care
Drug: IV Iron — Subjects will also receive IV iron per the FMCNA protocol that is standard of care at FMCNA clinics.

SUMMARY:
A phase 3b study for subjects receiving Epogen to compare a dosing algorithm between Hospira Epoetin and Standard of Care Epogen.

DETAILED DESCRIPTION:
Primary Objective: To evaluate switching from Epogen to Epoetin Hospira for maintenance of hemoglobin levels in anemic chronic kidney disease (CKD) subjects on hemodialysis using a specified algorithm for the dosing of erythropoietin stimulating agents (ESA).

Secondary Objective: To evaluate switching from Epogen to Epoetin Hospira on the dosing of ESA in anemic CKD subjects on hemodialysis using a specified algorithm for the dosing of ESA.

Exploratory Objectives: To generate hypotheses regarding maintenance of hemoglobin levels, dosing of ESA, intravenous (IV) iron dosing requirements, transferrin saturation (TSAT) levels and ferritin levels associated with the switch from Epogen to Epoetin Hospira in anemic CKD subjects on hemodialysis using specified algorithms for the dosing of ESA and for the dosing of IV iron, that are standard of care.

ELIGIBILITY:
Inclusion Criteria

Subjects eligible to be entered into the study will meet all of the following criteria:

1. Adult female or male subjects; age ≥ 18 years.
2. End stage renal disease subjects treated in-center with the modality of hemodialysis for ≥ 120 days.
3. Diagnosed with anemia.
4. Administered routine Epogen therapy for at least 16 weeks by an IV route for treatment of anemia using an Epogen version of an FMCNA dosing algorithm for ESA, and did not miss more than 3 prescribed doses of Epogen within 12 weeks prior to randomization.
5. Currently using the IV Epogen version of the ESA dosing algorithm cMAB 5 (inclusive of versions 5.0, 5.1, …) for anemia management.
6. Receiving hemodialysis at a clinic using the FMCNA dosing algorithm for IV iron that is the FMCNA standard of care treatment for iron replacement.

Exclusion Criteria

Subjects that meet any of the following criteria will be ineligible to be entered into the interventional cohort:

1. Subjects unable to provide a signed and dated informed consent for this clinical research study.
2. As determined by the Investigator, female subjects of child bearing potential who do not agree to use a highly effective method of contraception.
3. Any condition as determined by the investigator that would place a subject at an increased risk, or preclude subject's full compliance with the study procedures and visits.
4. Female subjects who are known to be or found to be, pregnant or lactating.
5. Subjects that are not a candidate for ESA therapies per the label warnings listed in the package insert for Epogen and/or contraindications to Epoetin Hospira listed in the Investigators' Brochure; or have had a known positive test for anti-rhEPO antibodies.
6. Treatment with any investigational drug within 30 days prior to randomization and throughout this clinical trial.
7. Diagnosed with any concurrent condition that could lead to greater-than-normal loss of blood, including but not limited to:

   * Menorrhagia, peptic ulcer disease, gastrointestinal bleeding, blood dyscrasia, hemoglobinopathy
   * Use of anticoagulation therapy, including warfarin with a target international normalized ratio (INR) of 2 or greater Anti-platelet therapy (e.g. aspirin or clopidogrel) is permitted, as is heparin given during hemodialysis. Low-dose warfarin is permitted and defined as the presence of at least two INR values less than or equal to 1.5 during the 120 days prior to enrollment and no values exceeding 1.5 at any time after 120 days prior to enrollment.

   Subjects started on warfarin with a known INR goal of 2.0 or greater are to receive no further treatment with the study drugs, but follow up visits can continue.

   Subjects on warfarin who meet criteria to enter the study are terminated if an INR > 2.0 is discovered or if no INR is available for 60 days.
8. History of transfusion of any blood product in the past 3 months, or 2 or more transfusions in the past 1 year; or donated or lost > 475 mL blood volume (including plasmapheresis) in the past 3 months.
9. Subjects currently receiving a long acting ESA, or who have received a long acting ESA in the 16 weeks prior to study randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 432 (Actual)
Dates: Start 2015-07-13 (Actual); Primary Completion 2016-07-02 (Actual); Study Completion 2016-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (44):
- United States (41):
  - California Institute of Renal Research, Chula Vista, California
  - California Institute of Renal Research at Fresenius Medical Care, Poway, California
  - Fresenius Medical Care Rancho, Rancho Bernardo, California
  - California Institute of Renal Research at Fresenius Medical Care Kearny Mesa, San Diego, California
  - Fresenius Medical Care Paradise Valley, San Diego, California
  - Fresenius Medical Care, Tampa, Florida
  - Genesis Clinical Research, LLC, Tampa, Florida
  - Frenova Renal Research, Boise, Idaho
  - Fresenius Medical Care North America - Liberty Dialysis, Boise, Idaho
  - Frenova Renal Research, Caldwell, Idaho
  - Fresenius Medical Care North America - Liberty Dialysis, Caldwell, Idaho
  - Frenova Renal Research, Meridian, Idaho
  - Fresenius Medical Care North America - Liberty Dialysis, Meridian, Idaho
  - Frenova Renal Research, Nampa, Idaho
  - Fresenius Medical Care North America - Liberty Dialysis, Nampa, Idaho
  - Fresenius Medical Care-Kalamazoo East, Kalamazoo, Michigan
  - Paragon Health PC DBA Nephrology Center, Kalamazoo, Michigan
  - Fresenius Medical Care-Oshtemo, Kalamazoo, Michigan
  - Fresenius Medical Care, Biloxi Dialysis Unit, Biloxi, Mississippi
  - North Gulfport, Gulfport, Mississippi
  - South Mississippi Kidney Center, Gulfport, Mississippi
  - FMC Charlotte, Charlotte, North Carolina
  - Metrolina Nephrology Associates, PA, Charlotte, North Carolina
  - Briggs Avenue Dialysis Center, Durham, North Carolina
  - Durham Nephrology Associates, Durham, North Carolina
  - FMC Matthews, Matthews, North Carolina
  - Fresenius Medical Care- Lansdale Dialysis, Lansdale, Pennsylvania
  - Delaware Valley Nephrology and Hypertension Associates, PC, Philadelphia, Pennsylvania
  - Fresenius Medical Care, Warwick, Rhode Island
  - Fresenius Crossville Dialysis Unit, Crossville, Tennessee
  - Fresenius Medical Care-Franklin, Franklin, Tennessee
  - Knoxville Kidney Center, PLLC, Knoxville, Tennessee
  - Fresenius Dialysis West, Knoxville, Tennessee
  - Nephrology Associates, PC, Nashville, Tennessee
  - Fresenius Medical Care - Austin North 4478, Austin, Texas
  - Research Management Inc, Austin, Texas
  - Mission Bend Dialysis (FMC#3971), Houston, Texas
  - Southwest Houston Research, Ltd., Houston, Texas
  - Gamma Medical Research Inc, McAllen, Texas
  - Rosenberg Dialysis (FMC#1197), Rosenberg, Texas
  - Fresenius Medical Care Weslaco, Weslaco, Texas
- Puerto Rico (3):
  - Fresenius Medical Care Carolina, Carolina
  - Fresenius Medical Care, Humacao
  - Fresenius Medical Care San Juan, San Juan

REFERENCES:
- [Derived] Chung EY, Palmer SC, Saglimbene VM, Craig JC, Tonelli M, Strippoli GF. Erythropoiesis-stimulating agents for anaemia in adults with chronic kidney disease: a network meta-analysis. Cochrane Database Syst Rev. 2023 Feb 13;2(2):CD010590. doi: 10.1002/14651858.CD010590.pub3. PMID 36791280
- [Derived] Thadhani R, Guilatco R, Hymes J, Maddux FW, Ahuja A. Switching from Epoetin Alfa (Epogen(R)) to Epoetin Alfa-Epbx (RetacritTM) Using a Specified Dosing Algorithm: A Randomized, Non-Inferiority Study in Adults on Hemodialysis. Am J Nephrol. 2018;48(3):214-224. doi: 10.1159/000492621. Epub 2018 Sep 7. PMID 30196301

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In this study, 432 participants were enrolled, however, only 418 participants were treated.
Groups:
- Epoetin Hospira: Participants received intravenous (IV) injection of Epoetin Hospira as per the analogous version of Fresenius Medical Care North America (FMCNA) Erythropoietin Stimulating Agent (ESA) dosing algorithm Corporate Medical Advisory board (cMAB algorithm 1) along with IV iron as per the FMCNA standard of care. Drug was administered up to maximum 3 times per week up to Week 24. Participants were followed up to Week 26.
- Epogen: Participants received their ongoing standard of care which included IV injection of Epogen, as per the current version of the FMCNA ESA dosing algorithm cMAB 5 along with IV iron as per the FMCNA standard of care. Drug was administered up to maximum 3 times per week up to Week 24. Participants were followed up to Week 26.
Period: Overall Study
Arm/Group | Epoetin Hospira | Epogen
Started | 212 | 206
Completed | 156 | 158
Not Completed | 56 | 48
Not completed — Adverse Event | 15 | 12
Not completed — Withdrawal by Subject | 7 | 1
Not completed — Protocol Violation | 27 | 26
Not completed — Physician Decision | 1 | 2
Not completed — Lost to Follow-up | 6 | 7

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all participants who received at least 1 dose of study medication after randomization into the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Epoetin Hospira | Epogen | Total
Number analyzed (Participants) | 212 | 206 | 418
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.5 (13.96) | 59.3 (14.23) | 59.9 (14.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 102 | 184
  Male | 130 | 104 | 234

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Time When Participants Had Hemoglobin Levels Between 9 to 11 Gram Per Deciliter (g/dL)
Time Frame: Week 17 up to Week 24
Population: FAS included all participants who received at least 1 dose of study medication after randomization into the study. Here, "Number of participants analyzed (N)" signifies those number of participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of Weeks
Arm/Group | Epoetin Hospira | Epogen
Number analyzed (Participants) | 178 | 173
Percentage of Weeks | 61.9330 [57.5106 to 66.1659] | 63.3305 [58.7061 to 67.7217]
Statistical Analysis 1: Comparison: Epoetin Hospira vs Epogen; Clustered binomial analysis using logistic regression method was performed and generalized estimating equation method was used to construct 95 percent (%) two-sided confidence intervals (CIs); Test type: Non-Inferiority or Equivalence — Non-inferiority was concluded since the lower bound of the 95% CI of the difference in percentage was greater than the non-inferiority margin (-12.5%); Difference in Percentage = -1.3975, 95% CI 2-sided [-7.6503 to 4.8553]

2. Secondary Outcome: Change From Baseline in Weekly Mean Study Medication Dose Over Final 8 Weeks of Study Treatment
Time Frame: Baseline (8 Weeks prior to randomization), Week 17 up to Week 24
Population: FAS included all participants who received at least 1 dose of study medication after randomization in to the study. Here, "N" signifies number of participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Units per week
Arm/Group | Epoetin Hospira | Epogen
Number analyzed (Participants) | 180 | 174
Units per week | -1861.8 (563.50) | -799.8 (573.14)
Statistical Analysis 1: Comparison: Epoetin Hospira vs Epogen; P-value was calculated using analysis of covariance (ANCOVA) model with treatment as factor and baseline ESA dose as covariate; Test type: Superiority or Other; p = 0.1874, ANCOVA; LS Mean Difference = -1062.0, 95% CI 2-sided [-2643.2 to 519.2], Standard Error of Mean 803.95

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as non serious in another participant, or one participant may have experienced both a serious and non serious event during the study.
Arm/Group | Epoetin Hospira | Epogen
Serious Adverse Events (participants affected / at risk) | 66/212 | 64/206
Other Adverse Events (participants affected / at risk) | 10/212 | 21/206
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Epoetin Hospira (N=212) | Epogen (N=206)
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 2 | 2
Angina pectoris (Cardiac disorders) | 0 | 1
Angina unstable (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 2 | 6
Cardiac failure congestive (Cardiac disorders) | 0 | 3
Cardio-respiratory arrest (Cardiac disorders) | 0 | 2
Coronary artery disease (Cardiac disorders) | 0 | 2
Diastolic dysfunction (Cardiac disorders) | 0 | 1
Hypertensive heart disease (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Hyperparathyroidism secondary (Endocrine disorders) | 1 | 0
Parathyroid disorder (Endocrine disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 2
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2
Asthenia (General disorders) | 0 | 1
Catheter site haemorrhage (General disorders) | 0 | 1
Chest discomfort (General disorders) | 1 | 0
Chest pain (General disorders) | 3 | 1
Condition aggravated (General disorders) | 4 | 3
Death (General disorders) | 2 | 0
Early satiety (General disorders) | 1 | 0
Generalised oedema (General disorders) | 0 | 1
Hernia (General disorders) | 0 | 1
Impaired healing (General disorders) | 0 | 2
Medical device site ulcer (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Systemic inflammatory response syndrome (General disorders) | 0 | 1
Ulcer haemorrhage (General disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Cellulitis of male external genital organ (Infections and infestations) | 0/130 | 1/104 — This event was gender specific.
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Device related sepsis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1
Endocarditis (Infections and infestations) | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 1
Graft infection (Infections and infestations) | 1 | 0
Incision site infection (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 2 | 0
Osteomyelitis (Infections and infestations) | 0 | 2
Osteomyelitis chronic (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 7 | 1
Pneumonia bacterial (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 2 | 0
Pyuria (Infections and infestations) | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 3 | 1
Septic shock (Infections and infestations) | 2 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 2
Wound infection (Infections and infestations) | 0 | 1
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 1 | 2
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Arteriovenous graft site haemorrhage (Injury, poisoning and procedural complications) | 1 | 1
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Intentional product misuse (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Post procedural pulmonary embolism (Injury, poisoning and procedural complications) | 0 | 1
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 1
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 2
Vascular access malfunction (Injury, poisoning and procedural complications) | 0 | 1
Vascular bypass dysfunction (Injury, poisoning and procedural complications) | 1 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Haemoglobin decreased (Investigations) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 4 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 5 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 1
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/130 | 0/104 — This event was gender specific.
Cerebrovascular accident (Nervous system disorders) | 2 | 1
Encephalopathy (Nervous system disorders) | 1 | 2
Hemiparesis (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 2 | 0
Syncope (Nervous system disorders) | 2 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0/82 | 1/102 — This event was gender specific.
Anxiety (Psychiatric disorders) | 1 | 0
Major depression (Psychiatric disorders) | 1 | 0
Obstructive uropathy (Renal and urinary disorders) | 1 | 0
Urethral haemorrhage (Renal and urinary disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Choking (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Tracheomalacia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0
Renal transplant (Surgical and medical procedures) | 1 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 1 | 2
Hypotension (Vascular disorders) | 0 | 2
Peripheral artery occlusion (Vascular disorders) | 0 | 1
Steal syndrome (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Epoetin Hospira (N=212) | Epogen (N=206)
Nausea (Gastrointestinal disorders) | 3 | 13
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.